CLINICAL TRIAL: NCT00852787
Title: Marinobufagenin as a Target for DIGIBIND in Hypertensive Patients With End-stage Renal Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: University of Toledo Health Science Campus (Other)
Responsible Party: Deepak Malhotra, MD, PhD, University of Toledo
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AG0115; 263-MA-707136-1
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2009-12

CONDITIONS: Hypertension; Hemodialysis
Keywords: Digoxin like substances; digibind; digoxin immune fab; end-stage-renal-disease; marinobufagenin
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic | interventions — digoxin antibodies Fab fragments

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low (Experimental): 0.1mg/kg
  Interventions: Drug: Digoxin immune fab
- Medium (Experimental): 0.4mg/kg
  Interventions: Drug: Digoxin immune fab
- High (Experimental): 1.6 mg/kg
  Interventions: Drug: Digoxin immune fab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Digoxin immune fab — Intravenously one time
  Other Names: Digibind
  Arms: High; Low; Medium
Drug: Placebo — Intravenously one time
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effects of the digibind drug on hemodialysis patients with high blood pressure. Digibind is used to treat toxicity from digoxin and digoxin-like molecules which may contribute to high blood pressure.

DETAILED DESCRIPTION:
High blood pressure is a very common problem in patients with kidney disease. Researchers have noted that there are certain molecules in the blood of these patients that may be contributing to the high blood pressure. In particular these molecules have been labeled as "digoxin-like substances." Digoxin is a drug made from a certain plant that may contribute to high blood pressure. In research animals with kidney failure, it has been noted that the use of Digibind helps to lower the blood pressure in these animals. Digibind is a drug made from sheep that is used to treat the toxicity from digoxin as well as toxicity from molecules similar to digoxin.

In this study, volunteers that are on hemodialysis and have high blood pressure will be given a placebo or the digibind drug intravenously on two separate visits. The volunteers will then wear a 24-hour blood pressure monitor and return the following day. Volunteers will receive the Digibind at one visit during the study, and the placebo on the other visit.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years of age
* On hemodialysis with predialysis BP > 150/90 but ≤ 180/110
* On at least one anti-hypertensive medication for 6 consecutive readings
* Able to have blood pressure measured in an arm
* Women of child bearing potential must not be pregnant; must use contraception during the study and for one month after the study
* Receiving adequate dialysis (KT/V > 1.2)
* Compliant with the dialysis schedule and duration

Exclusion Criteria:

* Pregnant or nursing women
* Arm blood pressure is not possible to obtain
* Currently on digitalis
* On any Digibind-type product in the past
* History of allergies to antibiotics
* History of asthma
* Medical or psychiatric disorders which are unstable or which might interfere with study assessments or safe participation in the study
* History of use of, or evidence of need for, digitalis-like products
* Inability to understand or provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-04; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | Screening, and 24-hour period after first infusion and after second infusion

SECONDARY OUTCOMES:
Marinobufagenin levels | Screening, and after first and second infusions

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Malhotra, MD, PhD, Principal Investigator — University of Toledo
Locations (1):
- University of Toledo Medical Center, Toledo, Ohio, United States

REFERENCES:
- [Background] Bagrov AY, Shapiro JI. Endogenous digitalis: pathophysiologic roles and therapeutic applications. Nat Clin Pract Nephrol. 2008 Jul;4(7):378-92. doi: 10.1038/ncpneph0848. Epub 2008 Jun 10. PMID 18542120
- [Background] Mohmand B, Malhotra DK, Shapiro JI. Uremic cardiomyopathy: role of circulating digitalis like substances. Front Biosci. 2005 Sep 1;10:2036-44. doi: 10.2741/1679. PMID 15970476
- [Background] Fedorova OV, Simbirtsev AS, Kolodkin NI, Kotov AY, Agalakova NI, Kashkin VA, Tapilskaya NI, Bzhelyansky A, Reznik VA, Frolova EV, Nikitina ER, Budny GV, Longo DL, Lakatta EG, Bagrov AY. Monoclonal antibody to an endogenous bufadienolide, marinobufagenin, reverses preeclampsia-induced Na/K-ATPase inhibition and lowers blood pressure in NaCl-sensitive hypertension. J Hypertens. 2008 Dec;26(12):2414-25. doi: 10.1097/HJH.0b013e328312c86a. PMID 19008721